CLINICAL TRIAL: NCT05344820
Title: The Effect of the Art-based Mandala Intervention on the Quality of Life of Cancer Patients Receiving Chemotherapy
Acronym: ARQULA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Principal Investigator, Elif Yıldırım Ayaz, Principal Investigator, Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ARQULA
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Cancer; Chemotherapy Effect; Fatigue; Quality of Life; Rumination; Alexithymia
Keywords: cancer; Chemotherapy Effect; Fatigue; Quality of Life; Rumination; Alexithymia
MeSH Terms: conditions — Neoplasms; Fatigue; Rumination Syndrome; Affective Symptoms

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mandala Intervention (Experimental): To the experimental group; Mandala practice will be done for 2 hours, once a week for 8 weeks.
  Interventions: Behavioral: Art based mandala
- Control (No Intervention): No intervention will be applied to the control group

INTERVENTIONS:
Behavioral: Art based mandala — To the experimental group; Mandala practice will be done for 2 hours, once a week for 8 weeks.
  Arms: Mandala Intervention

SUMMARY:
The aim of this study is to determine the effect of mandala application on fatigue, quality of life, rumination and alexithymia in cancer patients receiving chemotherapy.

DETAILED DESCRIPTION:
A randomized controlled study on the effect of mandala application on cancer related fatigue, quality of life, rumination and alexithymia in cancer patients receiving chemotherapy has not been found in the literature.

The aim of this study is to determine the effect of mandala application on fatigue, quality of life, rumination and alexithymia in cancer patients receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Conscious and no communication problems
* Being literate
* Having a cancer diagnosis
* Receiving chemotherapy treatment (planned to continue treatment for 8 more weeks)
* Willing to participate in our study voluntarily

Exclusion Criteria:

* Not being willing to participate in the research
* Desire to leave the study at any time
* Deterioration of compliance with the working criteria during the time of the study,
* Those who do not participate in up to four mandala applications during the study period
* Those who cannot use a pen
* Those with a diagnosis of psychiatric and neurological disease
* Patients who are scheduled for drug intervention, radiotherapy, surgery other than chemotherapy within 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
level of quality of life | 1 week
  Level of quality of life as assessed by the Quality of Life Scale for the Treatment and Research of Cancer (min:0, max:100,with higher values indicating a higher functioning in functional scales and an increased presence of symptoms in symptom scales)
level of fatigue | 1 week
  level of fatigue assessed by the Piper Fatigue Scale (min:0, max, 100, higher values means higher fatigue)

SECONDARY OUTCOMES:
level of alexithymia | 1 week
  level of alexithymia assessed by Toronto Alexythimia Scale (higher values means more alexithymic)
level of rumination | 1 week
  level of rumination assessed by ruminative thought scale (higher values means more ruminative thought)

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yıldırım Ayaz, M.D., Principal Investigator — Sultan Abdülhamid Training And Research Hospital
Locations (1):
- Sultan Abdülhamid Training and Research Hospital, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No